CLINICAL TRIAL: NCT06504706
Title: Effect of Matcha Tea Versus Green Tea on Salivary pH and Flow Rate in High Caries Risk Patients: A Randomized Controlled Trial
Brief Title: Effect of Matcha Tea Versus Green Tea on Salivary pH and Flow Rate in High Caries Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadier Mahmoud Ahmed Gad, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 28923
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Salivary pH
MeSH Terms: interventions — Tea

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: participants will be blinded to the type of tea they are drinking and investigators will be blinded as well
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Green Tea (Active Comparator): Green tea contains a significant amount of catechins, which are subgroup of flavonoids and play a vital role in maintaining health having strong bactericidal as well as antibacterial activity
  Interventions: Procedure: Green Tea
- Matcha Tea (Experimental): Matcha, powder of specially cultivated tea leaves, is gaining popularity in functional food and other food markets all over the world. Various studies have reported the difference in bioactive compounds in matcha as compared to green tea and other tea formulations
  Interventions: Procedure: Matcha Tea

INTERVENTIONS:
Procedure: Matcha Tea — Japanese tea rich in antioxidants and Catechins
  Arms: Matcha Tea
Procedure: Green Tea — Green tea rich in catechins
  Arms: Green Tea

SUMMARY:
Objectives: To evaluate the effect of green tea versus matcha tea on the salivary pH in high caries risk patients. Materials and methods: Total number of high caries risk patients were randomized into two equal groups (n=). Group 1 (intervention group) was given Matcha Tea and Group 2 (control group) was given green tea. A portable digital pH meter was used to measure the salivary pH at baseline and after consumption tea immediately, after 5 mins and after 10 mins.

DETAILED DESCRIPTION:
Study Settings:

The study will be carried out at the Conservative Dentistry Department, Faculty of Dentistry, Cairo University in Egypt. Ethical approval will be taken from the Research Ethics Committee of the faculty of Dentistry, Cairo University. Signed informed consent will be signed each participant.

Recruitment:

Participants will be recruited from the patients' flow at the clinics of the Conservative Dentistry Department of Faculty of Dentistry, Cairo university.

Materials:

The Commercially available green tea and matcha tea for this study will be Lipton Tea. For preparation of green tea, 2 gr of green tea will be poured into 150 mL boiling water (100°C), after 3 minutes, it will be ready for drinking. As well as for matcha tea, 3 gr of green tea will be poured into 150 mL hot water (70°C), after 3 minutes, it will be ready drinking(7) .

Methods:

On the study day, all subjects will be instructed to brush their teeth 45 minutes after eating breakfast. Between 9-11 a.m., saliva samples will be collected through spitting method, one hour after breakfast and 15 minutes after brushing(7)

. For making the subjects blind to which tea they are drinking, the prepared tea will be served in the dark glasses. After drinking the green tea and matcha tea, every subject will be asked to bend his head forward and spit his saliva into laboratory tube every 60 seconds for 2-5 minutes. Samples will be collected immediately and 5 minutes after drinking tea(7)

.

.

Aim of the study:

The aim of this study is to evaluate the effect of green tea versus matcha tea on the salivary pH in high caries risk patients.

Research question:

In high caries risk patients, will matcha tea have the same effect as green tea on salivary pH?

PICOTS:

P: High caries risk patients I: Matcha tea C: Green tea O: Salivary pH T: T1: baseline T2: immediately T3: 5 mins T4: 10 mins

ELIGIBILITY:
Inclusion Criteria:

-

1. High caries risk patients

1. Satisfactory cooperative behavior
2. Age between 20-45 years old
3. Males or females
4. Subjects who signed informed consent

Exclusion Criteria:

* 1. Systemic diseases 2. Drug consumption during 3 past months 3. Salivary gland disorders 4. History of radiotherapy 5. Smoking

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
salivary pH | baseline before administration of tea, immediately after administration of tea, 5 minutes after administration of tea and 10 minutes after administration of tea
  pH of saliva to be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No